CLINICAL TRIAL: NCT05348824
Title: Effect of Moringa Oleifera Leaf Extract Versus Sodium Hypochlorite as Root Canal Irrigant on Postoperative Pain and Bacterial Reduction in Mandibular Premolars With Necrotic Pulps: A Randomized Clinical Trial
Brief Title: Effect of Moringa Oleifera Leaf Extract on Postoperative Pain and Bacterial Reduction in Mandibular Premolars
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Alfred Loka, Principal Investigator (Endodontic Resident), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO 3 -7 -1
Record Dates: First submitted 2022-04-17; First posted 2022-04-27 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Necrotic Pulp
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moringa oleifera (Experimental)
  Interventions: Dietary Supplement: Moringa oleifera leaf
- Sodium hypochlorite (Active Comparator)
  Interventions: Drug: Sodium hypochlorite

INTERVENTIONS:
Dietary Supplement: Moringa oleifera leaf — Leaf extract preparation
  Arms: Moringa oleifera
Drug: Sodium hypochlorite — 2.5% sodium hypochlorite (household bleaching agent)
  Arms: Sodium hypochlorite

SUMMARY:
The aim of this study is to clinically compare the intensity of post-operative pain and the amount of bacterial reduction after using Moringa oleifera leaf extract solution during chemo-mechanical preparation, versus 2.5% NaOCl, in asymptomatic necrotic mandibular premolars treated in a single visit

ELIGIBILITY:
Inclusion Criteria:

1. Systematically healthy patient (ASA I,II).
2. Age between 20 and 55 years
3. Male or female.
4. Asymptomatic mandibular premolar teeth diagnosed with pulp necrosis with apical periodontitis.
5. Radiographic examination using Digora intraoral periapical sensor plate and software (Digora; Soredex, Helsinki, Finland) showing mandibular premolars with (smaller than 3 mm (0-2 mm)) periapical radiolucency.

Exclusion Criteria:

1. Medically compromised patients having significant systemic disorders. (ASA III or IV).
2. History of intolerance to NSAIDS.
3. Teeth with:

   * Immature roots
   * Vital pulp tissues.
   * Association with swelling.
   * Acute peri-apical abscess or acute exacerbation of a chronic abscess.
   * Mobility Grade II or III.
   * Previously accessed or endodontically treated
   * Deep periodontal pockets more than 4 mm
   * Vertical root fractures, coronal perforation, calcification, and external or internal root resorptions.
4. Patients who could not interpret the NRS.
5. Patients with diabetes, immune-compromising, and immunosuppression disease and pregnant women were, also, excluded.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | up to 48 hours postoperatively
  postoperative pain will be marked by the patient using the Numerical rating scale (NRS) chart which is an 11 point scale consisting of numbers from 0 through 10, where: 0: reading represents "no pain" 1-3: readings represent "mild pain" 4-6: readings represent "moderate pain" 7-10: readings represent "severe pain"

SECONDARY OUTCOMES:
Intracanal bacterial load change | First sample is taken at Time 0 "T0" then second sample taken after chemo-mechanical preparation on 15 minutes at Time 1 "T1".
  The intracanal bacterial load change will be determined using agar culture technique by counting the colony forming units per milliliter (CFUs/mL) before and after root canal preparation.